CLINICAL TRIAL: NCT00691054
Title: Phase II Trial of Abraxane® in the Treatment of Patients With Pancreatic Cancer Who Have Failed First-Line Treatment With Gemcitabine-Based Therapy
Brief Title: Abraxane Therapy in Patients With Pancreatic Cancer Who Failed First-Line Gemcitabine Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20080055; SCCC-2007096 (Other: UMiami Sylvester Comprehensive Cancer Center)
Record Dates: First submitted 2008-06-04; First posted 2008-06-05 (Estimated); Results first posted 2013-11-15 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-04

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abraxane (Experimental): One treatment-cycle is 28 days with chemotherapy (Abraxane® 100 mg/m2) given on day 1, 8, and 15, followed by rest on week 4.
  Interventions: Drug: Abraxane

INTERVENTIONS:
Drug: Abraxane — One treatment-cycle is 28 days with chemotherapy (Abraxane® 100 mg/m2) given on day 1, 8, and 15, followed by rest on week 4. Treatment cycles will be repeated every 28 days for as long as disease is not progressing and patient tolerates treatment
  Other Names: Paclitaxel Albumin-Stabilized Nanoparticle Formulation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well paclitaxel albumin-stabilized nanoparticle formulation works in treating patients with locally advanced or metastatic pancreatic cancer that did not respond to first-line therapy with gemcitabine.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish preliminary evidence of efficacy of paclitaxel albumin-stabilized nanoparticle formulation in patients with locally advanced (unresectable) or metastatic pancreatic cancer that failed first-line therapy with a gemcitabine hydrochloride-containing regimen.

Secondary

* To determine the safety and characterize the toxicity profile of this drug.
* To determine the complete, partial, and overall response rates and duration of response in patients with measurable disease.
* To determine CA 19-9 response.
* To determine progression-free survival.

OUTLINE: This is a multicenter study.

Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed, locally advanced (unresectable) or metastatic pancreatic cancer, and have failed first-line treatment with a gemcitabine-containing regimen.
2. Patients have to be 18 years-old or older
3. Able to give signed Informed consent
4. Adequate end-organ function with laboratory parameters as follows:

   * Neutrophils: 1.5 x10^9/L or greater
   * Plts: 100 x10^9/L or greater
   * Hemoglobin: ≥ 9.0g/dL
   * Serum Creatinine: ≤ 1.5mg/dL
   * Bilirubin: ≤ 1.5 times the upper limit of the normal range (ULN)
   * Alanine transaminase (ALT)/Aspartate transaminase (AST): ≤ 2.5 times ULN
5. Adequate contraception: For female (or male) patients, either post-menopausal, or for pre-menopausal surgically sterilized, or willing to use an acceptable method of birth control for the duration of the study
6. Measurable or non-measurable disease by RECIST criteria
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
8. Patients must be at least 3 weeks from prior therapies and must have recovered from prior toxicity
9. Life expectancy greater than 3 months
10. Willing and able to comply with the protocol requirement.
11. Patients must not have any peripheral neuropathy equal or greater than grade 2

Exclusion Criteria:

1. Chemotherapy within 3 weeks prior to enrollment
2. Radiation therapy or evidence of acute effects of radiation therapy within 2 weeks prior to enrollment.
3. Any major surgery within 4 weeks prior to enrollment
4. Peripheral neuropathy equal to or greater than grade 2
5. Clinical AIDS or known positive HIV serology
6. Evidence of concurrent, clinically evident malignancy, except inactive non-melanoma skin cancer and inactive cervical cancer diagnosed or other cancer for which the patient has been disease-free for five years
7. Unstable angina
8. New York Heart Association (NYHA) Grade II or greater congestive heart failure
9. History of myocardial infarction within 3 months
10. History of stroke within 3 months
11. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to enrollment, anticipation of need for major surgical procedure during the course of the study
12. Pregnant (positive pregnancy test) or lactating
13. Inability to comply with study and/or follow-up procedures
14. Participants with serious medical or psychiatric illness that would render chemotherapy unsafe are ineligible.
15. Participants cannot have been in another experimental drug study within 4 weeks of the first infusion of these study medications.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caio Max S. Rocha Lima, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center; Gilberto Lopes, MD, Principal Investigator — Johns Hopkins Singapore International Medical Centre
Locations (2):
- University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida, United States
- Johns Hopkins Singapore International Medical Centre, Singapore, Singapore

REFERENCES:
- [Result] Hosein PJ, de Lima Lopes G Jr, Pastorini VH, Gomez C, Macintyre J, Zayas G, Reis I, Montero AJ, Merchan JR, Rocha Lima CM. A phase II trial of nab-Paclitaxel as second-line therapy in patients with advanced pancreatic cancer. Am J Clin Oncol. 2013 Apr;36(2):151-6. doi: 10.1097/COC.0b013e3182436e8c. PMID 22307213

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abraxane
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Abraxane: Abraxane : One treatment-cycle is 28 days with chemotherapy (Abraxane® 100 mg/m2) given on day 1, 8, and 15, followed by rest on week 4. Treatment cycles will be repeated every 28 days for as long as disease is not progressing and patient tolerates treatment
Arm/Group | Abraxane
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: years] | 61 [24 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 20
Stage-IV Disease [Number; unit: participants] — Number of participants with stage IV disease at enrollment
  participants | 18

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Rate at 6 Months
Description: Overall survival was measured from the start of treatment (date of first dose of Abraxane® therapy) to date of death due to any cause. For patients who are alive, follow-up time will be censored at date of last contact.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abraxane
Number analyzed (Participants) | 19
percentage of participants | 58 [33 to 76]

2. Secondary Outcome: Number of Participants Showing Complete or Partial Response
Description: Number of participants showing complete or partial response to protocol therapy according to Response Evaluation Criteria In Solid Tumors(RECIST) v1.0 criteria for target lesions and assessed by CT/MRI. Per RECIST, Complete Response (CR) = Disappearance of all target lesions; Partial Response (PR), >= 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Abraxane
Number analyzed (Participants) | 19
participants | 1

3. Secondary Outcome: Number of Participants Showing Stable Disease
Description: Number of participants showing stable disease according to RECIST 1.0 criteria
Time Frame: 12 months
Measure: Number; unit: participants
Groups:
- Single Arm: Abraxane : One treatment-cycle is 28 days with chemotherapy (Abraxane® 100 mg/m2) given on day 1, 8, and 15, followed by rest on week 4. Treatment cycles will be repeated every 28 days for as long as disease is not progressing and patient tolerates treatment
Arm/Group | Single Arm
Number analyzed (Participants) | 19
participants | 6

4. Secondary Outcome: Progression-free Survival
Description: Median number of months participants experienced progression-free survival, according to Response Evaluation Criteria In Solid Tumors(RECIST) v1.0 criteria for target lesions and assessed by CT/MRI. Per RECIST, progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abraxane
Number analyzed (Participants) | 19
months | 1.7 [1.5 to 3.5]

5. Secondary Outcome: Number of Participants Experiencing Adverse Events
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Abraxane
Number analyzed (Participants) | 19
Participants | 19

6. Secondary Outcome: Median Overall Survival of Participants
Description: Median overall survival rate of participants measured in months
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abraxane
Number analyzed (Participants) | 19
months | 7.3 [2.8 to 15.8]

ADVERSE EVENTS:
Arm/Group | Abraxane
Serious Adverse Events (participants affected / at risk) | 10/19
Other Adverse Events (participants affected / at risk) | 12/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abraxane (N=19)
Grade 3-4 Neutropenia (Infections and infestations) | 6
Grade 3-4 Neutropenic Fever (Infections and infestations) | 2
Grade 3-4 Anemia (Blood and lymphatic system disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abraxane (N=19)
Grade 1-2 Nausea (Gastrointestinal disorders) | 12
Grade 1-2 Anorexia (Metabolism and nutrition disorders) | 9
Grade 1-2 Hypocalcemia (Metabolism and nutrition disorders) | 7
Grade 1-2 Vomiting (Gastrointestinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No